CLINICAL TRIAL: NCT01787474
Title: A Phase I/II Clinical Trial Testing the Safety and Feasibility of IL-21-Expanded Natural Killer Cells for the Induction of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Donor Natural Killer Cells in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0079; NCI-2014-00883 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2014-00841; 2012-0079 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NK cells) (Experimental): Patients receive filgrastim-sndz SC QD beginning on day -7 and continuing until ANC are equal or over 1000. Patients also receive fludarabine phosphate IV over 30 minutes and approximately 4 hours later followed by cytarabine IV over 1 hour on days -6 to -2 (days -6 to -3 for patients over age 60). Beginning 2-7 days after the last dose of fludarabine phosphate and cytarabine, patients receive membrane-bound interleukin-21-expanded haploidentical natural killer cells IV over 30 minutes thrice weekly for 3 doses over 4 days (Monday-Thursday only).
  Interventions: Drug: Cytarabine; Biological: Filgrastim; Biological: Filgrastim-sndz; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Membrane-bound Interleukin-21-Expanded Haploidentical Natural Killer Cells

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Membrane-bound Interleukin-21-Expanded Haploidentical Natural Killer Cells — Given IV
  Other Names: (mbIL21)-expanded Haploidentical NK Cells; mbIL21-expanded Haploidentical NK Cells

SUMMARY:
This phase I/II trial studies the side effects and best dose of donor natural kill cells and to see how well they work in treating patients with acute myeloid leukemia that does not respond to treatment (refractory) or has come back after a period of improvement (relapsed). Giving natural killer cells after high dose chemotherapy may boost the patient's immune system by helping it see the remaining cancer cells as not belonging in the patient's body and causing it to destroy them (called graft-versus-tumor effect).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety, feasibility, and maximum tolerated dose of membrane-bound interleukin 21 (mbIL21)-expanded haploidentical natural killer (NK) cells after induction chemotherapy with fludarabine (fludarabine phosphate), cytarabine, and filgrastim-sndz, Zarxio (filgrastim-sndz) (G-CSF) (FLAG).

SECONDARY OBJECTIVES:

I. Determine the persistence of adoptively-transferred expanded NK cells. II. Determine the immunophenotype and function of expanded NK cells. III. Determine the overall response of acute myeloid leukemia (AML) to this regimen.

IV. Correlate NK cell persistence, phenotype, and function with overall response.

V. Estimate the rate at which patients receiving this regimen are able to go to transplant.

OUTLINE: This is a phase I, dose-escalation study of membrane-bound interleukin-21-expanded haploidentical natural killer cells followed by a phase II study.

Patients receive filgrastim-sndz subcutaneously (SC) once daily (QD) beginning on day -7 and continuing until absolute neutrophil counts (ANC) are equal or over 1000. Patients also receive fludarabine phosphate intravenously (IV) over 30 minutes and approximately 4 hours later followed by cytarabine IV over 1 hour on days -6 to -2 (days -6 to -3 for patients over age 60). Beginning 2-7 days after the last dose of fludarabine phosphate and cytarabine, patients receive membrane-bound interleukin-21-expanded haploidentical natural killer cells IV over 30 minutes thrice weekly for 3 doses over 4 days (Monday-Thursday only).

After completion of study treatment, patients are followed up for 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or primary refractory AML; patients with relapsed AML after allogeneic stem cell transplantation, including those who have received donor lymphocyte infusions, are eligible if they have no active graft versus host disease (GVHD) and are off immunosuppression
* Have a haploidentical family peripheral blood donor selected for best possible killer cell immunoglobulin-like receptor (KIR) reactivity; KIR typing will not be indicated if there is only one haploidentical donor; KIR typing is advised to be done if feasible and does not delay transplant
* Karnofsky or Lansky performance scale (PS) greater or equal to 70
* Serum creatinine =< 2 mg/dl or creatinine clearance greater or equal than 40 cc/min; creatinine for pediatric patients =< 2 mg/dl or =< 2 times upper limit of normal for age (whichever is less)
* Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lungs for carbon monoxide (DLCO) >= 50% of expected, corrected for hemoglobin; for pediatric patients, if unable to perform pulmonary function tests (most children < 7 years of age), pulse oximetry >= 92% on room air by pulse oximetry
* Total bilirubin =< 2 mg/dl or =< 2.5 x upper limit of normal (ULN) for age (unless Gilbert's syndrome)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN for age
* Left ventricular ejection fraction >= 40%; no uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease
* Negative serum test to rule out pregnancy within 2 weeks prior to registration in females of childbearing potential (non-childbearing potential defined as premenarchal, greater than one year post-menopausal, or surgically sterilized)
* Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the investigator
* Negative serology for human immunodeficiency virus (HIV)
* DONOR: Donor must be 16 years of age or older and weigh at least 110 pounds
* DONOR: Donor must be a human leukocyte antigen (HLA)-haploidentical relative selected for best NK alloreactivity, defined as having a KIR gene present on the donor NK cells for which the relevant HLA haplotype (KIR ligand) is absent in the recipient and present in the donor or selected on the basis of activating KIR gene content
* DONOR: Donor must meet standard institutional eligibility and donor certification criteria for therapeutic cell product donation
* DONOR: Not be pregnant as defined by negative serum (beta human chorionic gonadotropin [beta HCG]) pregnancy test in females of childbearing potential (non-childbearing potential defined as premenarchal, previous surgical sterilization, or postmenopausal for > 12 months)
* DONOR: Evaluation: history and physical examination; laboratory examinations: hematology, electrolytes, chemistry; infectious disease screening and serology; HLA typing; KIR typing will not be indicated if there is only one haploidentical donor; KIR typing is advised to be done if feasible and does not delay transplant

Exclusion Criteria:

* Congestive heart failure < 6 months prior to screening
* Unstable angina pectoris < 6 months prior to screening
* Myocardial infarction < 6 months prior to screening
* Uncontrolled infection, defined as an infection which has not resolved spontaneously or does not show evidence of significant resolution after initiating appropriate therapy, excluding chronic asymptomatic viral infections (e.g., human papillomavirus [HPV], BK virus, hepatitis C virus [HCV], etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of natural killer (NK) cells, defined as the highest dose level at which no more than 2 patients in a 6-patient cohort experience a dose limiting toxicity during treatment | Day 28

SECONDARY OUTCOMES:
Complete remission rate (CR) | Day 56 following infusion of the NK cells
  Estimated with Kaplan-Meier estimator and tabulated with 95% confidence intervals. Cox proportional hazards regression will be used to model CR as a function of NK cell dose.
NK-cell numerical expansion in vivo defined as an absolute circulating donor-derived NK cell count that increases above the post-infusion level | Up to day 56
  Proportion of patients with successful in vivo NK-cell expansion estimated with a 95% confidence interval.
Time to transplantation (TTT) | Up to day 56
  Estimated with Kaplan-Meier estimator and tabulated with 95% confidence intervals. Cox proportional hazards regression will be used to model TTT as a function of NK cell dose.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Srour, MBCHB, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org